CLINICAL TRIAL: NCT07022782
Title: A Nutritional Intervention Based on the Principles of Mediterranean Diet as a Putative Regulator of Craving and Redox Status of Patients Under Medication-assisted Treatment With Methadone and Buprenorphine: The Study Protocol of a Randomized Controlled Trial (the MED-DOPE Study)
Brief Title: MEDiterranean Diet-driven Detoxification of OPioid Addicted patiEnts (MED-DOPE)
Acronym: MED-DOPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristidis Veskoukis (Other)
Collaborators: Organization Against Drugs (OKANA) (Unknown)
Responsible Party: Sponsor-Investigator, Aristidis Veskoukis, Assistant Professor, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 48383/3-2-2022
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Opioid Addiction
Keywords: Mediterranean diet; Opioid use disorders; Methadone; Buprenorphine; Oxidative stress; Antioxidants; Nutrition; Craving
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Nutrition (Experimental): The intevention group will comprise patients under medication-assisted treatment (MAT) who are active members of the therapeutic units of the Greek Organization Against Drugs (OKANA). The participants will be stratified into two subgroups, i.e., methadone maintenance treatment (MMT) and buprenorphine maintenance treatment (BMT), according to the maintenance treatment program they attend. The nutritional intervention based on the principles of Mediterranean diet will be administered to the participants of both MMT and BMT subgroups of the intervention group. The patients will consume meals three times (i.e., breakfast, lunch and dinner) per day for 90 days (i.e., three months).
  Interventions: Other: A nutritional intervention based on the principles of Mediterranean diet
- No intervention - Control group (No Intervention): The control group will comprise patients under medication-assisted treatment (MAT) who are active members of the therapeutic units of the Greek Organization Against Drugs (OKANA). The participants will be stratified into two subgroups, i.e., methadone maintenance treatment (MMT) and buprenorphine maintenance treatment (BMT), according to the maintenance treatment program they attend. No intervention wil be applied. The patients will follow their normal nutritional habbits.

INTERVENTIONS:
Other: A nutritional intervention based on the principles of Mediterranean diet — The patients will consume meals three times (i.e., breakfast, lunch and dinner) per day for 90 days (i.e., three months) that are based on the principles of Mediterranean diet.
  Arms: Intervention - Nutrition

SUMMARY:
The MED-DOPE (MEDiterranean diet-driven Detoxification of OPioid addicted patiEnts) study is a randomized controlled trial that aims to investigate the role of a nutritional intervention based on the principles of Mediterranean diet on craving, which is the primary outcome, and blood redox status of opioid-addicted patients under medication-assisted treatment with buprenorphine and methadone. In detail, the patients of the intervention group will consume three meals per day (i.e., breakfast, lunch and dinner) based on the principles of Mediterranean diet for 90 days. The patients of the control group will follow their normal nutritional habits. Craving as the primary outcome, quality of sleep and biochemical parameters such as blood redox status will be evaluated. It is hypothesized that the applied nutritional intervention will reduce craving, probably through the improvement of blood redox status, of the patients of the intervention group compared to the patients of the control group.

DETAILED DESCRIPTION:
Background: Methadone and buprenorphine are considered as the "gold standard" medication-assisted treatment (MAT) for patients with opioid use disorders (OUDs). Patients who suffer from OUDs usually experience serious health consequences in the psychosocial and the biochemical level. Specifically, they are at 10-fold higher mortality risk than those of the general population. Moreover, there are inconsistencies related to the efficacy of MAT (i.e., methadone and buprenorphine) on retention to treatment and opioid craving, that is a major psychosocial parameter to be improved towards successful rehabilitation. Craving is a central psychosocial component for addiction characterized by a strong urge to use an illicit substance that induces addiction. It appears that although MAT partially normalizes this parameter, patients with OUDs continue to experience craving for opioids leading to drug-seeking behavior and relapse. Furthermore, opioids such as heroine induce oxidative stress, a common toxic biochemical outcome. However, this is the case also for methadone and buprenorphine, although in a lower extent compared to heroine. Therefore, opioid-addiction induced oxidative stress seems to be rather neglected and needs further attention. Oxidative stress is a result of excessive reactive oxygen species generation, which may cause protein and lipid oxidation and oxidative modification of DNA. To that end, the use of plant-derived compounds as auxiliary therapeutic approaches, in combination with methadone and buprenorphine could be a promising approach towards enhancement of the effectiveness of MAT. The biological plausibility for the adoption of such a nutritional practice relies on the fact that plant components namely polyphenols exert potent antioxidant properties against oxidative stress. It has been clearly shown that pomegranate juice is such a physical product. A nutritional approach on the basis of Mediterranean diet could also be considered as an alternative approach towards rehabilitation from addiction to opioids. Indeed, Mediterranean diet has been associated with better health outcomes. Its beneficial effects on human health have largely been attributed to the antioxidant properties of its components, mainly polyphenols.

Objectives: The MED-DOPE (MEDiterranean diet-driven Detoxification of OPioid addicted patiEnts) study aims to investigate the role of a nutritional intervention based on the principles of Mediterranean diet on craving and blood redox status of patients with OUDs under buprenorphine and methadone. This diet scheme is rich in antioxidant compounds that, along with medication (i.e., methadone and buprenorphine), could putatively act beneficially on several health parameters of the patients with OUDs.

Methods: Three meals (i.e., breakfast, lunch and dinner) will be administered daily for 90 days to patients with OUDs under methadone and buprenorphine. In two time points namely Days 1 and 90 the patients will form the heroine craving questionnaire to assess craving, which is the primary outcome of MED-DOPE study. Blood samples will also be collected from the participants in order to measure redox biomarkers (i.e., glutathione concentration, total antioxidant capacity, concentraiton of protein carbonyls, glutathione reductase activity and glutathione peroxidase activity).

Anticipated Outcome: It is hypothesized that the applied nutritional intervention will reduce craving probably through the improvement of blood redox status.

Conclusion: MED-DOPE is a hypothesis-driven and evidence-based project that proposes a nutrition-based solution for craving amelioration in patients with OUDs under MAT, potentially assisting towards their successful rehabilitation and societal reintegration.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years of age
* Long-term heroine or other opioid drug use
* Suffering from physical and mental dependence due to chronic opioid use

Exclusion Criteria:

* Serious medical problems, such as infection by human immunodeficiency virus or hepatitis B virus
* Current use of anti-inflammatory medication
* Relapse to other addictive substances (i.e., opioids, methamphetamine, benzodiazepines, cannabis, tetrahydrocannabinol, amphetamine) - To rule out the use of such substances, all participants will undergo weekly urine tests during the three-month period of the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2025-08-18 (Estimated)

PRIMARY OUTCOMES:
Craving | Changes between Day 1 (pre) and Day 90 (post) will be assessed.
  The effects of the applied nutritional intervention on craving will be assessed through the Heroin Craving Questionnaire (HCQ), which is a validated self-reported instrument. It is consisted of 45 questions divided in 5 dimensions, namely desire to use heroine, intentions and planning to use heroine, anticipation of positive outcome, relief from withdrawal or dysphoria, and lack of control overuse. The score is calculated with a 7-point Likert scale ranging from 1 (i.e., strongly disagree) to 7 (i.e., strongly agree) and the higher the score, the worse the outcome. HCQ will be completed by the volunteers of both the experimental and control groups at two timepoints as follows: Before the start of the experiment (i.e., Day 1 or pre) and at the end of the experiment (i.e., day 90 or post).

SECONDARY OUTCOMES:
Quality of Sleep | Changes between Day 1 (pre) and Day 90 (post) will be assessed.
  Quality of sleep of the patients will be assessed through the Pittsburgh Sleep Quality Index (PSQI), which is a 19-item self-reported questionnaire. It subjectively assesses sleep quality and quantity, sleep habits related to quality and occurrence of sleep disturbances in adults. It is consisted by 7 components, each of which has a score that is marked on a 0-3-Likert scale. Finally, the PSQI is calculated as the sum of the 7 components ranging between 0 and 21. Higher obtained scores indicate increased sleep complaints and lower sleep quality.
Blood GSH concentration | Changes in GSH concentration will be compared between Day 1 (pre) and Day 90 (post).
  The concentration of reduced form of glutathione (GSH) as a crucial intrinsic antioxidant metabolite will be measured spectrophotometrically in erythrocytes.
Concentration of protein carbonyls in blood | Changes in protein carbonyl concentration will be compared between Day 1 (pre) and Day 90 (post).
  The concentration of protein carbonyls, as a biomarker of protein oxidation, will be evaluated spectrophotometrically in plasma.
Total antioxidant capacity of blood | Changes in TAC will be compared between Day 1 (pre) and Day 90 (post).
  Total antioxidant capacity (TAC) will be evaluated spectrophotometrically in plasma.
Activity of glutathione reductase | Changes in glutathione reductase activity will be compared between Day 1 (pre) and Day 90 (post).
  The activity of glutathione reductase as an antioxidant enzyme will be measured in erythrocytes.
Activity of glutathione peroxidase | Changes in glutathione peroxidase activity will be compared between Day 1 (pre) and Day 90 (post).
  The activity of glutathione peroxidase as an antioxidant enzyme will be measured in erythrocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Christonikos Leventelis, Principal Investigator — Organization Against Drugs (OKANA)
Locations (1):
- Organization Against Drugs (OKANA), Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this investigation will be provided, upon request respecting GDPR, to qualified researchers and clinicians with related academic interest.

REFERENCES:
- [Background] Veskoukis AS, Tsatsakis AM, Kouretas D. Dietary oxidative stress and antioxidant defense with an emphasis on plant extract administration. Cell Stress Chaperones. 2012 Jan;17(1):11-21. doi: 10.1007/s12192-011-0293-3. Epub 2011 Sep 30. PMID 21956695
- [Background] Leventelis C, Makri S, Ververi A, Papageorgiou K, Tentolouri A, Mountzouridi E, Tekos F, Barmpas PT, Tasoulis S, Metsios GS, Kouretas D, Veskoukis AS. Pomegranate juice ameliorates craving and oxidative stress on patients under medication for opioid addiction treatment with methadone and buprenorphine: A ranzomised controlled trial. Clin Nutr ESPEN. 2025 Apr;66:34-45. doi: 10.1016/j.clnesp.2025.01.025. Epub 2025 Jan 10. PMID 39798867
- [Background] Leventelis C, Goutzourelas N, Kortsinidou A, Spanidis Y, Toulia G, Kampitsi A, Tsitsimpikou C, Stagos D, Veskoukis AS, Kouretas D. Buprenorphine and Methadone as Opioid Maintenance Treatments for Heroin-Addicted Patients Induce Oxidative Stress in Blood. Oxid Med Cell Longev. 2019 Apr 9;2019:9417048. doi: 10.1155/2019/9417048. eCollection 2019. PMID 31093318
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Billingsley HE, Carbone S. The antioxidant potential of the Mediterranean diet in patients at high cardiovascular risk: an in-depth review of the PREDIMED. Nutr Diabetes. 2018 Mar 9;8(1):13. doi: 10.1038/s41387-018-0025-1. PMID 29549354
- [Background] Arezoomandan M, Zhiani R, Mehrzad J, Motavalizadehkakhky A, Eshrati S, Arezoomandan R. Inflammatory, oxidative stress and cognitive functions in patients under maintenance treatment with methadone or buprenorphine and healthy subjects. J Clin Neurosci. 2022 Jul;101:57-62. doi: 10.1016/j.jocn.2022.04.018. Epub 2022 May 6. PMID 35533613
- [Background] Aleksandrova K, Koelman L, Rodrigues CE. Dietary patterns and biomarkers of oxidative stress and inflammation: A systematic review of observational and intervention studies. Redox Biol. 2021 Jun;42:101869. doi: 10.1016/j.redox.2021.101869. Epub 2021 Jan 22. PMID 33541846